CLINICAL TRIAL: NCT06002880
Title: Clinical Evaluation of OBU When Used for Indirect Dental Restorations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: Kerr Corporation (Industry)
Responsible Party: Principal Investigator, Sibel Antonson, Professor and Assistant Dean for Research and Development, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kerr 04-2022
Record Dates: First submitted 2023-07-24; First posted 2023-08-21 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (8):
- Post/Core-Total Etch (Experimental): Endodontic posts and/or cores-Total etch
  Interventions: Device: Optibond Universal
- Ceramic-Total Etch (Experimental): Glass-ceramics-Total etch
  Interventions: Device: Optibond Universal
- Metal/Zi-Total Etch (Experimental): Metal-Zi-Total etch
  Interventions: Device: Optibond Universal
- Composite-Total Etch (Experimental): Composite-Total etch
  Interventions: Device: Optibond Universal
- Post/Core-Self Etch (Experimental): Endodontic posts and/or cores-Self etch
  Interventions: Device: Optibond Universal
- Ceramic-Self Etch (Experimental): Glass-ceramics-Self etch
  Interventions: Device: Optibond Universal
- Metal/Zi-Self Etch (Experimental): Metal-Zi-Self etch
  Interventions: Device: Optibond Universal
- Composite-Self Etch (Experimental): Composite-Self etch
  Interventions: Device: Optibond Universal

INTERVENTIONS:
Device: Optibond Universal — OBU™ will be used used for the cementation of indirect restorations (ceramic restorations, composite, zirconia and metal crowns) and pretreatment for indirect restoration, according to manufacturer's Instruction For Use in self-etch and total-etch modes.

SUMMARY:
The objective of this study is to evaluate the clinical safety and performance of Optibond Universal (OBU), a single component universal dental adhesive intended for indirect dental restorations according to manufacturer's Instruction For Use.

DETAILED DESCRIPTION:
The device used in the study, Optibond Universal (OBU) is a single component universal dental adhesive intended for direct and indirect dental restorations. OBU is formulated to provide reliable bond strength with any etch technique, on all common substrates and in combination with any resin cement without auxiliary products (silane or metal primers) even in absence of light. OBU is intended for general population use by a dental professional.

OBU contains an acidic component to etch the tooth surface in order to allow the adhesive to mechanically adhere to the prepared tooth surface. The adhesive can be used with light or without light cured prior to application of the restorative material. This allows for the adhesive to mechanically and chemically bond to the applied restorative material. OBU is formulated to provide a reliable bond strength, and it's compatible with all etching modes (self-etch, selective etch, and total etch).

Aim/Hypothesis/Objective The primary objective of this study is to evaluate the clinical performance of OBU used in the intended clinical conditions.

The device will undergo evaluation in the following categories:

Functional Properties Endodontic posts Ceramic restorations Composite and metal crowns Pretreatment for indirect restorations Core build-ups

Endpoints:

Primary endpoints:

Evaluation of clinical safety and performance of OBU, a single component universal dental adhesive intended for indirect dental restorations according to manufacturer's Instruction For Use.

(Indirect metal restoration is defined as any restoration made of precious or non-precious alloy such as inlays, onlays, porcelain fused to metal, metal full coverage crown, metal full coverage fixed partial denture). All implant restorations are excluded.

Secondary endpoints:

Post-operative sensitivity, retention, general periodontal health, and general optical properties after baseline, 6 months, 1 year and 2 years post-placement.

The hypothesis to be tested is that OBU is safe and effective in clinical settings when the device is used according to manufacturer's instructions:

H0: P ̂_T-P ̂_C≥ ∆ HA: P ̂_T-P ̂_C< ∆ Where ∆ (delta) refers to the non-inferiority margin set at 10%.

ELIGIBILITY:
Inclusion Criteria:

* Is willing to provide voluntary written informed consent in English.
* Is in good medical health and able to tolerate the dental procedures.
* Has 1 qualifying either vital or endodontically treated molar and/or premolar that requires an endodontic post and or core build-ups with subsequent indirect restoration or an indirect restoration only. Only 1 tooth per quadrant can be included in the study if more than 1 tooth in need of restoration. The maximum number of restorations will not exceed two per patient.
* The tooth must be restorable, i.e. without subgingival caries and must have a minimum of 2-3 mm healthy supragingival tooth structure.
* Study teeth must have an antagonist in the opposite jaw and have a neighboring tooth on at least one side.
* Study teeth must be vital and without any symptoms suggesting irreversible damage of the pulp, or endodontically treated and hermetically filled according to standards of care (i.e., free of clinical signs and symptoms of periapical pathology).

Exclusion Criteria:

* Is currently taking part in an evaluation of other dental procedures.
* Has chronic periodontitis or rampant caries.
* The study tooth exhibits clinical signs of periapical pathology.
* The study tooth has a history of self-reported preoperative pulpal problems.
* The study tooth that has been restored using eugenol containing materials.
* Study Subjects with severe parafunctional habits or occlusal issues affecting the subject teeth.
* Women who are pregnant (self-reported). It is standard of care to postpone routine dental procedures and radiographed until after pregnancy.
* Women who are breast feeding.
* Known allergy to methacrylates or other components of resin composites, local anesthetics, or metals used for dental restorations.
* An employee of the sponsor or members of their immediate family.
* Condition affecting salivary flow (e.g., salivary gland disorder, Sjögren's Syndrome, xerogenic medications).
* Are unwilling or unable to have dental radiographs or photographs taken of their dentition and soft tissues.
* Unable to return to the recall visits.
* Any other condition which is the view of the investigator may affect the ability of a patient to complete the study.
* Teeth with implant restorations.
* Third molars.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity Questionnaire-Visual Analog Scale 0 to 10 (0=No pain, 10=Worst pain possible) | Screening
  Preoperative sensitivity
Sensitivity Questionnaire-Visual Analog Scale 0 to 10 (0=No pain, 10=Worst pain possible) | Preparation, Provisional Restoration (up to 6 weeks from Screening)
  Preoperative sensitivity
Sensitivity Questionnaire-Visual Analog Scale 0 to 10 (0=No pain, 10=Worst pain possible) | 48 hours after Cementation (up to 4 weeks from Preparation)
  Postoperative sensitivity
Sensitivity Questionnaire-Visual Analog Scale 1 to 5 (1=No pain, 5=Worst pain possible) | Baseline Followup Assessments (approximately 3 weeks from Cementation)
  Postoperative sensitivity
Sensitivity Questionnaire-Visual Analog Scale 1 to 5 (1=No pain, 5=Worst pain possible) | 6-months Followup Assessments (approximately 6 months from Baseline)
  Postoperative sensitivity
Sensitivity Questionnaire-Visual Analog Scale 1 to 5 (1=No pain, 5=Worst pain possible) | 1-year Followup Assessments (approximately 1 year from Baseline)
  Postoperative sensitivity
Sensitivity Questionnaire-Visual Analog Scale 1 to 5 (1=No pain, 5=Worst pain possible) | 2-Year Followup Assessments (approximately 2 years from Baseline)
  Postoperative sensitivity
FDI (World Dental Federation) Clinical Evaluation Criteria-Modified | Baseline Followup Assessments
  Functional Properties, Biological Properties, Aesthetic Properties (1 clinically excellent-5 clinically poor Scale)
FDI (World Dental Federation) Clinical Evaluation Criteria-Modified | 6-months Followup Assessments
  Functional Properties, Biological Properties, Aesthetic Properties (1 clinically excellent-5 clinically poor Scale)
FDI (World Dental Federation) Clinical Evaluation Criteria-Modified | 1-year Followup Assessments
  Functional Properties, Biological Properties, Aesthetic Properties (1 clinically excellent-5 clinically poor Scale)
FDI (World Dental Federation) Clinical Evaluation Criteria-Modified | 2-Year Followup Assessments
  Functional Properties, Biological Properties, Aesthetic Properties (1 clinically excellent-5 clinically poor Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Antonson, Principal Investigator — NSU CDM
Locations (1):
- Nova Southeastern University, College of dental Medicine, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill EE. Dental cements for definitive luting: a review and practical clinical considerations. Dent Clin North Am. 2007 Jul;51(3):643-58, vi. doi: 10.1016/j.cden.2007.04.002. PMID 17586148
- [Background] Alharbi A, Rocca GT, Dietschi D, Krejci I. Semidirect composite onlay with cavity sealing: a review of clinical procedures. J Esthet Restor Dent. 2014 Mar-Apr;26(2):97-106. doi: 10.1111/jerd.12067. Epub 2013 Dec 17. PMID 24341472
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774